CLINICAL TRIAL: NCT04660422
Title: Advance Care Planning: Communicating With Outpatients for Vital Informed Decisions
Brief Title: Advance Care Planning: Communicating With Outpatients for Vital Informed Decision
Acronym: ACP-COVID
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, James A. Tulsky, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 20-600; UH3AG060626-03S1 (NIH)
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Advanced Care Planning; Shared Decision Making; Video Decision Aids; Communication Skills; Advance Directives; Natural Language Processing; Covid19
Keywords: Covid 19; Advanced Care Planning; Shared decision making; Video decision aids; Communication skills; Serious illness decision making; Health care proxy; Advance directives; Natural language processing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-COVID-19 ACP baseline: Two six-month control periods prior to the wide-scale implementation of the intervention, allow us to measure a baseline rate of ACP activity and identify the "pre-COVID-19 ACP baseline rate" and a "COVID-19 ACP baseline rate.
  September 15, 2019 - March 14, 2020,
  Interventions: Other: Medical Record Review
- COVID-19 rate: Two six-month control periods prior to the wide-scale implementation of the intervention, allow us to measure a baseline rate of ACP activity and identify the "pre-COVID-19 ACP baseline rate" and a "COVID-19 ACP baseline rate.
  March 15, 2020 - September 14, 2020
  Interventions: Other: Medical Record Review
- ACP rate: ACP rate during the implementation period, which begins December 15, 2020 and continues for six months, to the rates in the previous two control periods December 15, 2020-June 15, 2021
  Interventions: Other: VitalTalk communication skills training; Other: ACP Decisions Video Program; Other: Intervention training:; Other: Medical Record Review

INTERVENTIONS:
Other: VitalTalk communication skills training — Clinicians will receive VitalTalk intensive communication skills training via highly structured Zoom conference. They will learn skills relevant to discussions about ACP and COVID-19 including delivering serious news, eliciting goals of care, and managing difficult conversations via telehealth platforms.
  Groups: ACP rate
Other: ACP Decisions Video Program — All clinicians will also be trained remotely on the ACP Decisions Video Program using the ACP app. Training will instruct clinicians on how to: 1. Introduce the COVID-19 videos to patients and caregivers; 2. Select the appropriate video(s) from the entire suite according to patients' needs; and, 3. Prescribe videos for patients and caregivers using the electronic platform. The suite of ACP videos is designed to address common ACP decisions confronting patients at risk or with COVID-19 and the caregivers.
  Groups: ACP rate
Other: Intervention training: — Training will instruct the clinicians on how to: i. more effectively communicate with patients regarding COVID- 19, ii. have ACP conversations with patients, iii. introduce the videos to patients and families, iv. use the videos as an adjunct to ACP counseling by clinicians, v. select the appropriate video(s) from the entire suite as according to patients' needs, and, vi. use the app or electronic platform for prescribing videos to be seen at home (telehealth visits), or to be viewed in clinic with an iPad.
  Groups: ACP rate
Other: Medical Record Review — 13,000 (total) patients aged 65 or older for our primary (completed advance care plans) outcome. ACP can include designating a health care proxy, discussion of advance directives, goals-of-care discussions, CPR discussions, palliative care discussions and referrals, as well as hospice. Each of these ACP outcomes will also be compared in secondary analyses using NLP. These data will be obtained from the EHR. All patient participants will only be included for medical record review.

SUMMARY:
This Pre-Post, open-cohort design, pragmatic trial with 150 clinicians and will evaluate the effectiveness of the use of telehealth Advanced Care Planning (ACP) Program by comparing ACP documentation among 13,000 patients over 65

DETAILED DESCRIPTION:
This study is investigating if the use of telehealth ACP Program will improve and sustain rates of ACP from the time that the intervention is implemented compared to two time periods prior to the intervention. The Comprehensive ACP Program combines two widely disseminated interventions to assess impact when used concurrently.

* One is VitalTalk clinician communication skills training (www.vitaltalk.org) during which the primary care clinicians will practice ACP with simulated patient actors under the guidance of a trained VitalTalk facilitator.
* The second is the ACP Decisions video decision aids (www.acpdecisions.org) which are directed to patients and provide education about ACP. This inclusive ACP approach treats patients and clinicians as equal stakeholders providing both with the communication skills and tools needed to make decisions about COVID-19 medical care before the toughest choices arise.
* The training is four cumulative hours, most of which is spent in communication skills work, and the remainder learning how to introduce the videos into one's practice. No patients participate in the training. The ambulatory practices included in this intervention gain access to the ACP Decisions videos, which can be introduced to patients. Videos may be seen in clinic or sent to patients' homes via an electronic or paper code.
* We will recruit up to 30 clinicians from participating clinics who completed the intervention training and ask them to complete a qualitative interview to learn about their experience with the ACP intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinic Eligibility: Clinics affiliated with Northwell Health may be included in the study.
* Clinician, Staff Eligibility: Any staff member identified by the site-PIs are affiliated with Northwell Health.
* Patient Eligibility: To be eligible for this study, individuals must be aged 65 or over, affiliated with the Northwell Health clinic. For each of the three periods of the study, those patients over the age of 65 who are engaged (e.g., seen in person, telehealth, etc.) with the clinic during that time period will be included in that time period

Exclusion Criteria:

* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: To be eligible for this study, individuals must be aged 65 or over, affiliated with the Northwell Health clinic. For each of the three periods of the study, those patients over the age of 65 who are engaged (e.g., seen in person, telehealth, etc.) with the clinic during that time period will be included in that time period.
Sampling Method: Non-Probability Sample
Enrollment: 42019 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rate for Advanced Care Planning (ACP) documentation | 2 Years
  This study tests the effects of an ACP Program that trains clinicians and provides patients with a video decision aid on rates of ACP among 13,000 patients at risk, or with, COVID-19. All patients over 65 engaged with the enrolled clinics over the course of each time period in each of the three study periods will be included in the analysis. Rates of ACP are determined by natural language processing data extraction of electronic health records. Generalized linear mixed models will be used to compare outcomes between intervention and control periods.

SECONDARY OUTCOMES:
Rate of orders for resuscitation preferences | 2 years
  Same methodology as Primary Outcome
Rate of palliative care consultation | 2 years
  Same methodology as Primary Outcome
Rate of referral to hospice | 2 years
  Same methodology as Primary Outcome
Advanced Care Planning (ACP) documentation rates among under-represented minority groups. | 2 Years
  The analysis will use a difference in differences approach comparing the changes from the control period to the intervention period between White and non-White racial minority and between non-Medicaid and Medicaid patients.

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tulsky, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Northwell Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Murray GF, Lakin JR, Paasche-Orlow MK, Tulsky JA, Volandes A, Davis AD, Zupanc SN, Carney MT, Burns E, Martins-Welch D, LaVine N, Itty JE, Fix GM. Structural Barriers to Well-grounded Advance Care Planning for the Seriously Ill: a Qualitative Study of Clinicians' and Administrators' Experiences During a Pragmatic Trial. J Gen Intern Med. 2023 Dec;38(16):3558-3565. doi: 10.1007/s11606-023-08320-2. Epub 2023 Jul 24. PMID 37488368
- [Derived] Volandes AE, Zupanc SN, Paasche-Orlow MK, Lakin JR, Chang Y, Burns EA, LaVine NA, Carney MT, Martins-Welch D, Emmert K, Itty JE, Moseley ET, Davis AD, El-Jawahri A, Gundersen DA, Fix GM, Yacoub AM, Schwartz P, Gabry-Kalikow S, Garde C, Fischer J, Henault L, Burgess L, Goldman J, Kwok A, Singh N, Alvarez Suarez AL, Gromova V, Jacome S, Tulsky JA, Lindvall C. Association of an Advance Care Planning Video and Communication Intervention With Documentation of Advance Care Planning Among Older Adults: A Nonrandomized Controlled Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220354. doi: 10.1001/jamanetworkopen.2022.0354. PMID 35201306